CLINICAL TRIAL: NCT04518397
Title: Sankofa Paradigm: A Healing-centered, Therapeutic Theatre Program for Girls Ages 7 -18
Brief Title: Sankofa Paradigm: A Therapeutic Theatre Program for Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Boys & Girls Clubs of Indianapolis (Unknown); Community Health Network (Other)
Responsible Party: Principal Investigator, Sally Wasmuth, Assistant Professor Occupational Therapy, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: The Sankofa Paradigm
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-05

CONDITIONS: Adolescent Behavior; Child Behavior; Mental Health Wellness 1; Mental Health Wellness 2
MeSH Terms: conditions — Adolescent Behavior; Child Behavior

STUDY DESIGN:
Intervention Model Description: Pre/post cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theatre participants (Experimental): Girls in this arm will participate in the theatre intervention.
  Interventions: Behavioral: Theatre

INTERVENTIONS:
Behavioral: Theatre — 6-week participatory arts culturally-informed theatre program

SUMMARY:
The purpose of this study is to test the impact of a 6-week theatre intervention rooted in African culture (Sankofa) on the wellness of girls (predominately African American) ages 8-18 receiving services at five Boys & Girls Club Indianapolis sites. Theatre interventions are led by Asante theatre personnel and evaluated by the PI and occupational therapy graduate students. The theatre intervention being evaluated has been conducted for decades by an established theatre company with widespread community participation and anecdotal positive responses, but has not been scientifically evaluated to understand how it impacts wellbeing. This will be the first large-scale study of the mechanisms of change and of the impact of the theatre intervention in the community and will help to guide future therapeutic interventions using theatre with underserved populations.

Research questions include: Is Sankofa a feasible and acceptable intervention for the target population? Does participation in Sankofa result in improved scores on wellness outcome measures, including the National Youth Outcomes Initiative (NYOI) survey?

The study is funded by Asante Children's Theatre via the Central Indiana Community Foundation Women's Fund.

DETAILED DESCRIPTION:
This project will take place over a 3 year period and will consist of 10 6-week theatre interventions (5 for girls 8-12 and 5 for girls 13-18). The first two (pilot) interventions (one for each age group) are scheduled to take place in Spring of 2020. From Fall 2020 through Spring 2022, one intervention per age group will be implemented each fall and one per age group each spring.

The theatre intervention is an Asante Theatre production that involves reading a script, being assigned a role, rehearsing, participating in discussions about the script that will contribute to script development/editing to personalize it, and eventually performing the play in front of a community audience. The play is free and open to the public and at the end of the performance participants will participate in a community conversation during which audience members can ask questions about the process. The talk back is moderated by the PI, and participants are not required to respond to questions but can speak up if/when they feel comfortable doing so. Theatre interventions are led by Asante theatre personnel and evaluated by the PI and occupational therapy graduate students. Evaluations take place after the PI obtains parental/guardian informed consent, the week after the intervention, 6 weeks follow up, and 6 months follow up. Evaluation sessions are conducted individually with each girl who signs up to participate, using data collection tools described below and attached in the 'notes/attachment' section, and will take no longer than 60 minutes. Adult audience members at performances are also participants of this study if they consent by checking "Yes" or "No" on the Audience Survey and responding to questions. The audience survey is described briefly below and attached in the notes/attachments section.

For 4 weeks leading up to each intervention, recruit will take place through posting flyers throughout the Boys & Girls Club of Indianapolis (BGCI) where the interventions are to take place (implemented at 5 different clubs throughout the city). Flyers will also be circulated through BGCI social media and listservs, and sent home to parents. Girls who want to participate can let BGCI staff members know and BGCI staff will provide that girl's parent/guardian with an informed consent document to review and sign with the PI's contact information on it in case the parent/guardian has questions. The PI will call parents to ensure understanding and answer questions. She will also review the document to obtain assent from girls who want to participate and have their parents' signed consent forms.

ELIGIBILITY:
Inclusion Criteria:

* Female identifying
* Member of Boys and Girls Club of Indianapolis

Ages: 7 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 163 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
National Youth Outcomes Initiative | baseline, 6-weeks, compared to national average
  change in leadership, competence, and social and emotional development; 45 Likert-type items; 43 scored 1-4 scale, 2 items scored on 1-5 scale, higher scores indicate better outcomes. Max score of 182.

CONTACTS AND LOCATIONS:
Locations (1):
- Finish Line Boys and Girls Club, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No